CLINICAL TRIAL: NCT03397147
Title: Pilot Sleep Intervention to Improve Diabetes Management in School-Aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Jaser, Associate Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 171902
Record Dates: First submitted 2018-01-02; First posted 2018-01-11 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Randomized trial with 2 conditions (intervention and usual care).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual Care
- Sleep Coach Jr. (Experimental): Parents randomized to the intervention condition will receive a binder with the treatment manual, and the intervention will be administered in person (first session) and via telephone (second session) on an individual basis. The first session will focus on parent education and developing a positive bedtime routines, and the second session will be used to address barriers specific to the individual child.
  Interventions: Behavioral: Sleep Coach Jr.

INTERVENTIONS:
Behavioral: Sleep Coach Jr. — A brief sleep education program for parents of school-aged children with type 1 diabetes, with a focus on resolving sleep disturbances with parent education and positive bedtime routines.
  Arms: Sleep Coach Jr.

SUMMARY:
Evaluate the feasibility, acceptability, and preliminary efficacy of a sleep-promoting intervention for school-aged children with type 1 diabetes and their caregivers in a pilot randomized trial. The primary outcome is improvements in child sleep, and secondary outcomes include glycemic control (HbA1c, % in range), improvements in parent sleep, parental distress, and child behavior problems.

ELIGIBILITY:
Inclusion Criteria:

* child between 5-9 years of age
* child have been diagnosed with type 1 diabetes for at least 12 months
* caregiver lives with child
* caregiver can read/speak English

Exclusion Criteria:

* child has other major health problems or sleep disorders other than insufficient sleep or insomnia
* participating in other intervention studies

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Child Sleep Duration | 3 months
  Child sleep duration (measured with actigraphy)
Child Sleep Quality | 3 months
  Child sleep quality (measured with Child Sleep Habits Questionnaire)

SECONDARY OUTCOMES:
Glycemic Control | 3 months
  HbA1c, % glucose values in range
Parent Sleep Duration | 3 months
  Parent sleep duration (measured with actigraphy)
Parental Well-being | 3 months
  Well-Being Index (World Health Organization Five Well-Being Index, WHO-5)
Child Behavior Problems | 3 months
  Behavior problems measured with the Child Behavior Checklist (CBCL)
Parent Sleep Quality | 3 months
  and sleep quality (measured with Pittsburgh Sleep Quality Index)
Parental Fear of Hypoglycemia | 3 months
  Parental fear of hypoglycemia (Hypoglycemic Fear Survey, Worry subscale)
Parental Diabetes Distress | 3 months
  Diabetes distress (Problem Area In Diabetes - Parental Version Revised)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States